CLINICAL TRIAL: NCT00205179
Title: Alzheimer's Disease: Potential Benefit of Isoflavones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-048; 5K23AG024302-03 (NIH); A534255 (Other: University of Wisconsin, Madison); SMPH/MEDICINE/MEDICINE*G (Other: University of Wisconsin, Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Novasoy treated (Experimental): 100mg/day soy isoflavones
  Interventions: Drug: Novasoy
- Placebo (Placebo Comparator): 100mg/day matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Novasoy — 100mg/day soy isoflavones
  Arms: Novasoy treated
Drug: Placebo — 100mg/day matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this pilot study is to evaluate the potential effects of soy isoflavone supplements on cognitive function for men and women with Alzheimer's Disease (AD). Preliminary studies evaluating the effects of soy supplements on memory in cognitively healthy older adults have yielded promising results that are now being evaluated in patients with AD. It is hypothesized that isoflavone supplements will ameliorate cognitive declines for older adults diagnosed with Alzheimer's disease, when compared to subjects on placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD
* Has reliable and available caregiver to assist with medication and appointments
* On a stable dose of cholinesterase inhibitor, or if unable to tolerate medication, patient has no plans to re-initiate cholinergic therapies while in the study

Exclusion Criteria:

* Current or recent use (<6 months) of menopausal Hormone Replacement Therapy (HRT)
* Current or recent use (<4 months) or oral antibiotic therapy
* Typical dietary intake of soy isoflavones >5 mg/day
* History or significant gastro-intestinal or colon disease, or colon/intestinal resection
* Irritable bowel syndrome
* History of breast cancer, or abnormal mammogram within 12 months
* History of chronic obstructive pulmonary disease, diabetes mellitus, liver disease or unstable ischemic heart disease
* Significant neurological disease other than AD that might affect cognitive function, such as stroke, Parkinson's disease, multiple sclerosis, or serious traumatic brain injury

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey E Gleason, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Result] Gleason CE, Carlsson CM, Barnet JH, Meade SA, Setchell KD, Atwood CS, Johnson SC, Ries ML, Asthana S. A preliminary study of the safety, feasibility and cognitive efficacy of soy isoflavone supplements in older men and women. Age Ageing. 2009 Jan;38(1):86-93. doi: 10.1093/ageing/afn227. Epub 2008 Dec 2. PMID 19054783
- [Result] Gleason CE, Fischer BL, Dowling NM, Setchell KD, Atwood CS, Carlsson CM, Asthana S. Cognitive Effects of Soy Isoflavones in Patients with Alzheimer's Disease. J Alzheimers Dis. 2015;47(4):1009-19. doi: 10.3233/JAD-142958. PMID 26401779

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 subjects withdrew consent; 3 subjects ineligible due to abnormal laboratory tests or inability to complete testing
Period: Overall Study
Arm/Group | Novasoy | Placebo
Started | 32 | 33
Completed | 30 | 29
Not Completed | 2 | 4
Not completed — Death | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Older adults with Alzheimer's disease
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Novasoy | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.8 (6.8) | 75.7 (7.7) | 76 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33 | 31 | 64
  Latino | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 33 | 32 | 65
Number of participants with Apolipoprotein E4 (ApoE4) allele [Count of Participants; unit: Participants] — One subject in each group declined to undergo ApoE genotyping Population: One subject in each group declined to undergo ApoE genotyping
  Participants
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 15 | 16 | 31
Education in years [Mean (Standard Deviation); unit: years] | 14.2 (2.5) | 14.8 (2.7) | 14.5 (2.6)
Total weekly isoflavone intake at Baseline [Mean (Standard Deviation); unit: mg/week] — Established with Food Frequency Questionnaire (FFQ)
  mg/week | 6.5 (34.1) | 16.5 (66.3) | 12.5 (45.2)
Global cognition: Mini-Mental State Examination score [Mean (Standard Deviation); unit: score on a scale] | 22.4 (5.3) | 23.5 (4.0) | 22.95 (4.65)
Mood symptoms: Geriatric Depression Scale-Short Form score [Mean (Standard Deviation); unit: score on scale] | 2.6 (2.4) | 3.2 (3.3) | 2.9 (2.85)
Number of participants on Acetylcholinesterase-Inhibitors (AchE-I) [Count of Participants; unit: Participants] — Acetylcholinesterase-Inhibitors included Donepezil, Galantamine Hydrobromide, and Rivastigmine4NMDA-
  Participants | 30 | 31 | 61
Number of participants on N-methyl-D-aspartate receptor (NMDAR) blocker-Memantine [Count of Participants; unit: Participants] | 14 | 16 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (5.4) | 27.5 (5.0) | 27.7 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Outcomes - Language Executive Function : Category Fluency Assessed as Number of Words Generated/Min
Description: Participants are given 1 min to produce as many unique words as possible within a category (category fluency). More words per minute will correlates to better category fluency
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of words generated per minute
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 27
number of words generated per minute | 21.5 (1.9) | 25.7 (2.0)

2. Primary Outcome: Cognitive Outcomes - Language Executive Function : Phonemic Fluency/Verbal Fluency Assessed as Number of Words Generated Per Minute
Description: Participants are given 1 min to produce as many words as possible starting with a given letter (letter fluency). More number of words per minute correlates to better phonemic fluency/verbal fluency
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of words generated per minute
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 28
number of words generated per minute | 25.9 (2.4) | 35.2 (2.4)

3. Primary Outcome: Immediate and Delayed Recall on Verbal Memory/ List Learning Immediate and Delayed Free Recall: Number of Words Recalled
Description: List of 15 semantically unrelated words is presented verbally to the participants once, after which they are asked to free recall as many words as possible. Subsequently, this presentation-test routine (learning trials) is repeated four more times. A total recall score is determined by adding the number of recalled items for the five learning trials. After presentation of a distractor list and a delay of approximately 20 minutes, participants are asked to freely recall items from the original word list. A delayed recall score is then derived from this test.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of words recalled
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 29 | 28
Number of words recalled | 1.8 (0.50) | 2.2 (0.50)

4. Primary Outcome: Immediate and Delayed Recall on Verbal Memory/ Logical Memory Immediate and Delayed Recall: Number of Story Elements Recalled
Description: In the logical delayed memory test, participants are read a logically organized story. Approximately 20 minutes later, the participants are asked to recall the story from memory (Delayed Recall). The version used in this study uses only one story (Story A) read once to participants at each study visit. Possible scores for delayed recall trials range from 0 to 25, with higher scores reflecting more details recalled.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of story elements recalled
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 29 | 28
Number of story elements recalled | 4.6 (0.95) | 5.7 (0.9)

5. Primary Outcome: Measure of Divided Attention: Time to Complete Trail Making Test B
Description: Trail Making Test-Version B (TMT B) [113], a measure of divided attention, the subject is asked to draw lines to connect consecutively numbered and lettered circles, alternating between the 2 sequences. The time needed to complete the task is recorded.
  More time taken to complete the test or higher score indicates lower executive function/higher impairment.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 25 | 27
Seconds | 95.5 (16.7) | 95.7 (16.0)

6. Primary Outcome: A Test of Planning: Time to Complete Mazes
Description: Time to complete mazes is a test of planning. Subjects are asked to complete a set of 3 mazes. The time taken to complete the maze is inversely proportional to the cognitive function.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 27 | 26
Seconds | 32.2 (5.3) | 22.6 (5.4)

7. Primary Outcome: Measure of Selective Attention: Time to Complete Stroop Color Word Test
Description: Selective attention was evaluated with the Stroop Color Word Interference Test. In the interference portion of this test, the subject identifies the color of ink in which words ("red", "green", or "blue") are printed, requiring the subject to inhibit their natural tendency to read the word. A subject's score is the time taken to identify 50 stimulus items.
  The time taken to complete the maze is inversely proportional to the cognitive function.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 27 | 27
Seconds | 105 (12) | 91.8 (12)

8. Primary Outcome: Visual Memory Test: Complex Figure Delayed Recall; Number of Points
Description: Visual memory will be evaluated by complex figure delayed recall test. In this test , a two dimensional figure is shown to the subjects. After a delay of 30 min, they are asked to draw the same figure based on their memory. The Complex Figure Test assesses the subject's ability to remember a 2-dimensional figure presented briefly. The scoring system used includes scores related to location, accuracy and organization. Higher score correlates to better visual memory.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of points
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 29
number of points | 10.6 (1.8) | 13.4 (1.8)

9. Primary Outcome: Visual Memory : Benton Visual Retention Test: Number of Correct Figures
Description: The Benton Visual Retention Test (or simply Benton test or BVRT) is an individually administered test for people aged from 8 years to adulthood that measures visual perception and visual memory. It can also be used to help identify possible learning disabilities among other afflictions that might affect an individual's memory. The individual examined is shown 10 designs, one at a time, and asked to reproduce each one as exactly as possible on plain paper from memory. The test is untimed, and the results are professionally scored by form, shape, pattern, and arrangement on the paper.
  For the 'test of number of correct figures' score is calculated based on an all-or-nothing approach; points are awarded if the reproduction of the design matches the original.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of correct figures
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 28
number of correct figures | 2.7 (0.4) | 2.8 (0.4)

10. Primary Outcome: Cognitive Outcomes - Visual Memory : Benton Visual Retention; Number of Errors
Description: The Benton Visual Retention Test is an individually administered test for people aged from 8 years to adulthood that measures visual perception and visual memory. It can also be used to help identify possible learning disabilities among other afflictions that might affect an individual's memory. The individual examined is shown 10 designs, one at a time, and asked to reproduce each one as exactly as possible on plain paper from memory. The test is untimed, and the results are professionally scored by form, shape, pattern, and arrangement on the paper.
  For the 'test of number of errors' score is calculated based on the number and type of errors made for each design. The major categories for these errors are omissions, distortions, perseverations, rotations, misplacements, and size errors.These scores are then be compared to several sets of normative data available in the manual, each representing different demographic characteristics, and conclusions can be drawn by the examiner.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of errors
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 28
Number of errors | 14.5 (1.2) | 13.1 (1.2)

11. Secondary Outcome: Cognitive Outcomes - Visual Motor : Complex Figure Copy; Number of Points
Description: Visual memory will be evaluated by Complex Figure copy test. The Complex Figure Test assesses the subject's ability to copy a 2-dimensional figure. The scoring system used include scores related to location, accuracy and organization. Higher score correlates to better visual memory.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: number of points
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 28 | 29
number of points | 27.6 (1.1) | 29.0 (1.1)

12. Secondary Outcome: Cognitive Outcomes - Visual Motor : Time to Complete Grooved Pegboard Test Using the Dominant Hand
Description: The Grooved Pegboard is a dexterity test consisting of 25 holes with randomly positioned slots. Pegs with a key on one side must be rotated to match the hole before they can be inserted. Participants are instructed to place all pegs into the 25 holes, picking up one at a time, and using just one hand. They use their dominant hand. Time taken to finish the test inversely correlates to the cognitive ability.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: time in seconds
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 24 | 27
time in seconds | 134.3 (17.6) | 149.8 (16.6)

13. Secondary Outcome: Cognitive Outcomes - Visual Motor : Time to Complete Grooved Pegboard Test Using the Non-Dominant Hand
Description: The Grooved Pegboard is a dexterity test consisting of 25 holes with randomly positioned slots. Pegs with a key on one side must be rotated to match the hole before they can be inserted. Participants are instructed to place all pegs into the 25 holes, picking up one at a time, and using just one hand. They use their non-dominant hand. Time taken to finish the test inversely correlates to the cognitive ability.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: time in seconds
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 22 | 26
time in seconds | 161.8 (24.4) | 156 (22.4)

14. Secondary Outcome: Cognitive Outcomes-Global Cognition : Mini-Mental State Examination (MMSE) Score
Description: During the MMSE, a health professional asks a participant a series of questions designed to test memory, ability to solve simple problems and other thinking skills.
  The maximum MMSE score - 30 points. Score of 20 to 24 - mild dementia, 13 to 20 - moderate dementia, and <12 indicates severe dementia.
  On average, the MMSE score of a person with Alzheimer's declines about 2 to 4 points each year.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 29 | 30
score on a scale | 21.3 (1.0) | 23.4 (1.0)

15. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Depression Scale
Description: Depression scale is one of the subscale of POMS. Depression scale has 15 items and scores ranges from 0-60. Higher score indicates more severe depression.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 9 (1.8) | 11.4 (1.7)

16. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Tension Scale
Description: Tension scale is one of the subscale of POMS. Tension scale has 9 items and scores ranges from 0-36. Higher score indicates more severe outcomes.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 8.2 (1.3) | 9.3 (1.3)

17. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Anger Scale
Description: Anger scale is one of the subscale of POMS. Tension scale has 12 items and scores ranges from 0-48. Higher score indicates more anger issues.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 6.8 (1.4) | 8.3 (1.4)

18. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Fatigue Scale
Description: Fatigue scale is one of the subscale of POMS. Tension scale has 7 items and scores ranges from 0-28. Higher score indicates more fatigue.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 10.3 (1.2) | 10.3 (1.2)

19. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Vigor Scale
Description: Vigor scale is one of the subscale of POMS. Vigor scale has 8 items and scores ranges from 0-32. Higher score indicates more severe outcomes.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 12.4 (1.1) | 12.0 (1.1)

20. Secondary Outcome: Multiple Mood States: Profile of Mood States (POMS)-Confusion Scale
Description: Confusion scale is one of the subscale of POMS. Confusion scale has 7 items and scores ranges from 0-28. Higher score indicates more severe outcomes.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 28 | 28
score on a scale | 15.5 (1.1) | 14 (1.1)

21. Secondary Outcome: Geriatric Depression Scale-Subject Report
Description: Geriatric Depression Scale (GDS) has been tested and used extensively with the older population to measure depression.
  Subject will self-report a short form GDS consisting of 15 questions. Out of 15 items, 10 indicate the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicate depression when answered negatively.
  Scores of 0-4 are considered normal, depending on age, education, and complaints; Scores of 5-8 indicate mild depression; 9-11 indicate moderate depression; and Scores of 12-15 indicate severe depression.
  The Short Form is more easily used by physically ill and mildly to moderately demented patients who have short attention spans and/or feel easily fatigued. It takes about 5 to 7 minutes to complete
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 29 | 28
score on a scale | 2.1 (0.6) | 3.3 (0.6)

22. Secondary Outcome: Geriatric Depression Scale-Study Partner Report
Description: Study partner is someone who has frequent contact with the subject (e.g. an average of 10 hours per week or more), and can accompany the subject to all clinic visits for the duration of the protocol.
  Study partner will report a short form GDS consisting of 15 questions. Out of 15 items, 10 indicate the presence of depression when answered positively, while the rest (question numbers 1, 5, 7, 11, 13) indicate depression when answered negatively.
  Scores of 0-4 are considered normal, depending on age, education, and complaints; Scores of 5-8 indicate mild depression; 9-11 indicate moderate depression; and Scores of 12-15 indicate severe depression.
  The Short Form is more easily used by physically ill and mildly to moderately demented patients who have short attention spans and/or feel easily fatigued. It takes about 5 to 7 minutes to complete.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 29 | 28
score on a scale | 5.2 (0.7) | 6.3 (0.7)

23. Secondary Outcome: Number of Participants With ApoE4 Allele
Description: The epsilon-4 allele of the apolipoprotein E gene (APOE4) has been consistently associated with a greater risk of Alzheimer's disease (AD) as well as an earlier onset of AD.
  Determination of apolipoprotein E (APOE) genotype was performed on a non-fasting blood sample collected at Baseline, using standard Polymerase chain reaction (PCR) and DNA sequencing techniques in a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory. DNA extracted from whole blood was amplified by PCR using specific primers for the ApoE gene and the DNA then sequenced and analyzed for genotype using the FinchTV program (Version 1.3; Geospiza, Inc.)
Time Frame: Baseline
Population: Older adults with Alzheimer's disease
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Novasoy
Number analyzed (Participants) | 33 | 32
Participants | 15 | 16

24. Secondary Outcome: Plasma Concentrations of Isoflavones at Baseline
Description: Isoflavone assays will be performed on non-fasting blood samples collected at baseline.
  Novasoy capsules predominantly contain purified glycoside forms of isoflavones known genistein and diadzein. The plasma level of genistein and diadzine will be measured in the participants plasma.There is large inter-individual variations in the extent of intestinal metabolism, even when the quantity of isoflavone intake is standardized. Equol is a metabolite of isoflavones. Equol has high biological efficacy. Therefore, along with genistein and diadzein, plasma levels of equol will be measured to understand the isoflavone metabolism in the participants.
Time Frame: baseline
Population: Data is unavailable for 2 subject from placebo group and 1 subjects from Novasoy group
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 33 | 32
ng/ml
  Genistein: number analyzed (Participants) | 31 | 31
  Genistein | 4.8 (11.4) | 1.5 (2.6)
  Daidzein | 2.8 (6.1) | 1.3 (2.5)
  Equol | 0.3 (1.5) | 0.1 (0.5)

25. Secondary Outcome: Plasma Concentrations of Isoflavones at Month 3
Description: Isoflavone assays will be performed on non-fasting blood samples collected at month 3.
  Novasoy capsules predominantly contain purified glycoside forms of isoflavones known genistein and diadzein. The plasma level of genistein and diadzine will be measured in the participants plasma.There is large inter-individual variations in the extent of intestinal metabolism, even when the quantity of isoflavone intake is standardized. Equol is a metabolite of isoflavones. Equol has high biological efficacy. Therefore, along with genistein and diadzein, plasma levels of equol will be measured to understand the isoflavone metabolism in the participants.
Time Frame: At month 3
Population: Data is unavailable for 1 subject from each group
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 33 | 32
ng/ml
  Genistein: number analyzed (Participants) | 32 | 31
  Genistein | 2.1 (3.7) | 2777.7 (188.4)
  Daidzein | 1.1 (2.3) | 197.3 (150.5)
  Equol | 0.2 (0.5) | 20.3 (50.7)

26. Secondary Outcome: Plasma Concentrations of Isoflavones at Month 6
Description: Isoflavone assays will be performed on non-fasting blood samples collected at month 6.
  Novasoy capsules predominantly contain purified glycoside forms of isoflavones known genistein and diadzein. The plasma level of genistein and diadzine will be measured in the participants plasma.There is large inter-individual variations in the extent of intestinal metabolism, even when the quantity of isoflavone intake is standardized. Equol is a metabolite of isoflavones. Equol has high biological efficacy. Therefore, along with genistein and diadzein, plasma levels of equol will be measured to understand the isoflavone metabolism in the participants.
Time Frame: At month 6
Population: Data is unavailable for 1 subject from placebo group and 3 subjects from Novasoy group
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 33 | 32
ng/ml
  Genistein: number analyzed (Participants) | 32 | 29
  Genistein | 15.6 (35.4) | 338.6 (308.8)
  Daidzein | 10.6 (37.8) | 206.6 (156.8)
  Equol | 0.1 (0.6) | 19.6 (40.5)

27. Secondary Outcome: Plasma Concentrations of Estradiol at Baseline
Description: Estradiol assay will be performed on non-fasting blood samples collected at baseline using an enzyme immunoassay kit.
Time Frame: baseline
Population: Estradiol analysis done by the same investigator as part of another project with different subjects (PMID: 9054783 linked in the citation), did not show any change in the estradiol levels. Based on that, investigators did not see the justification for running these analyses in the current study. No estradiol analyses were performed for this study.
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Plasma Concentrations of Estradiol at 3 Month
Description: Estradiol assay will be performed on non-fasting blood samples collected at baseline using an enzyme immunoassay kit.
Time Frame: At 3 month
Population: as for outcome 27
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Plasma Concentrations of Estradiol at 6 Month
Description: Estradiol assay will be performed on non-fasting blood samples collected at baseline using an enzyme immunoassay kit.
Time Frame: At 6 month
Population: as for outcome 27
Arm/Group | Placebo | Novasoy Treated
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Active: 100mg/day soy isoflavones
  Novasoy: 100mg/day soy isoflavones
Arm/Group | Active | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 3/33
Other Adverse Events (participants affected / at risk) | 25/32 | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=32) | Placebo (N=33)
Death (Nervous system disorders) | 0 (0) | 2 (2) — Death due to complications from Alzheimer's disease
Seizures (Nervous system disorders) | 1 (1) | 0 (0) — Developed seizures secondary to Alzheimer's
DVT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=32) | Placebo (N=33)
other illness not related to treatment (General disorders) | 25 (25) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No